CLINICAL TRIAL: NCT01847183
Title: Evaluation of an Intranet-Based Alcohol Prevention Program in Middle School
Brief Title: Evaluation of an School-based Alcohol Prevention Program for Middle School Students
Acronym: AlcoholINET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA019671; R01AA019671 (NIH)
Record Dates: First submitted 2013-04-25; First posted 2013-05-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol-related Disorders; Drinking and Driving; Neurological Impairment
Keywords: heavy drinking; prevention; high school; adolescence
MeSH Terms: conditions — Alcohol-Related Disorders; Driving Under the Influence; Neurologic Manifestations | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Click City®: Alcohol (Experimental): Receive the Click City®: Alcohol program as part of their school curriculum.
  Interventions: Behavioral: Click City®: Alcohol
- Usual Curriculum (No Intervention): Students receive their usual alcohol curriculum

INTERVENTIONS:
Behavioral: Click City®: Alcohol — A school based program, Click City®: Alcohol consists of 12 effective components delivered in 7th grade and a booster of 5 effective components delivered in 8th grade.
  Arms: Click City®: Alcohol

SUMMARY:
The purpose of this research is to create and evaluate the efficacy of an exciting (fun to use), and potentially disseminable computer-based prevention program, Click City®: Alcohol, for use by 7th graders with a booster in 8th grade students. The ultimate goal of Click City®: Alcohol is to prevent the onset of heavy drinking during high school and post-high school. Secondary goals of the program include decreasing students' intentions and willingness to engage in heavy drinking in high school. The proposed program is unique both in its delivery system and the development process.

Aim 1: The investigators plan to develop and test approximately 24 components over the first two years of the study.

Aim 2: The final Click City®: Alcohol program will consist of 12 effective components delivered in six sessions over a three-week period in 7th grade. This is followed by two booster sessions, consisting of a total of 5 components delivered over a one-week period in 8th grade. Educational newsletters to parents and teacher guides will accompany the program.

Aim 3: Following development, the investigators will conduct a group randomized trial to evaluate the efficacy of this program as compared to schools' usual alcohol prevention curriculum. The investigators plan to recruit, stratify and randomly assign 26 middle schools to one of the two conditions, Click City®: Alcohol and Usual Curriculum (UC). Students in the Click City®: Alcohol and yoked UC schools will be assessed prior to the beginning of the 7th grade program, following the 7th grade program, following the 8th grade booster, which would occur approximately one year after the 7th grade program, and a follow-up assessment in the 9th grade to assess long-term outcomes, one year after the 8th grade assessment.

DETAILED DESCRIPTION:
The proposed program is unique both in its delivery system and the development process. The program will be delivered in a computer game like format over a school-based intranet system (i.e., networked computers linked to a school-based server), which enables users to interact individually with the program and to share their experiences by receiving immediate feedback on both their own responses and those of their classmates' collective responses. The delivery of this computer-based programs assures fidelity of implementation. Each activity (component) ultimately included in the program will be continually developed and tested to assure that it is effective at changing the targeted theoretically based etiological mechanism (risk factor). Development will include an experimental assessment to evaluate the effectiveness of each component and only effective components will be included in the program. The 7th grade version of Click City®: Alcohol program will consist of 12 effective components delivered in six sessions over a three-week period. This will be followed by two 8th grade booster sessions, consisting of a total of 5 components delivered over a one-week period. Educational newsletters to parents and teacher guides will be developed to accompany the program. The investigators will conduct a randomized efficacy trial with 26 middle schools. Half of the schools will use the newly developed program and the other half will use the programs that they usually do to teach about Alcohol.

ELIGIBILITY:
Inclusion Criteria:

* parents give passive consent for their students to participate. Students must attend a participating school.

Exclusion Criteria:

* non-English speakers, some special Ed students

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2300 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Decrease intentions to get drunk from baseline to one week follow-up; from baseline to one-year follow-up and from baseline to two-year followup. | one week following intervention; one year following intervention: two years following intervention
  Intention is measured by two items:
  Do you think you will get drunk (from drinking too much alcohol) when you are in high school? Do you think you will get drunk (from drinking too much alcohol) when you are older?

SECONDARY OUTCOMES:
Decrease willingness to get drink alcohol from baseline | one week following intervention; one year following intervention: two years following intervention
  Willingness is measured by:
  This is a "suppose" question. Think about yourself in this situation. We are not saying that you would be in this situation. We just want you to think about it, then tell us how you would act. Suppose you were with a group of friends and there was some alcohol there and you could have it if you wanted. How willing would you be to do each of the following:
  (check on Not at all willing, a little willing, kind of willing, pretty willing, very willing)
  1. Drink one drink
  2. Drink more than one drink
  3. Drink enough to get buzzed
  4. Drink enough to get drunk

CONTACTS AND LOCATIONS:
Overall Officials: Judy Andrews, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States